CLINICAL TRIAL: NCT02315014
Title: Effect of Balanced Daily Protein Distribution Supplemented With Whey Protein on Muscle Protein Synthesis in Overweight Older Men During Calorie Restriction and Exercise (ARC III)
Brief Title: Daily Protein Intake Distribution and MPS (ARCIII)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12.12.NRC
Record Dates: First submitted 2014-11-13; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- whey protein (Experimental): whey protein micelles
  Interventions: Other: whey protein
- placebo (Placebo Comparator): calorie-free placebo
  Interventions: Other: placebo

INTERVENTIONS:
Other: whey protein — whey protein.
  Arms: whey protein
Other: placebo — placebo.
  Arms: placebo

SUMMARY:
To determine whether a balanced total daily dietary protein distribution supplemented with whey protein during a weight-loss intervention will result in increased muscle protein synthesis

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI 27-40 kg/m2)
* Non-smokers
* Non-diabetic
* No history of hyperlipidemia
* Not taking medications thought to interfere with study
* Considered generally healthy

Exclusion Criteria:

* Efforts to lose weight in previous 16 weeks
* Hyperlipidemia
* Blood pressure ≥ 140/90 mmHg
* Smoking
* Heart and other organ disease
* Type 2 diabetes
* Gastrointestinal disease
* Orthopedic injury interfering with exercise
* Use of certain medications (HRT, antihypertensives, diuretics, antiarythmia medications, antiresorptive agents, anabolic agents, hypoglycemic agents, and statins known to affect muscle i.e. Simvastatin and Zocor)

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
muscle protein synthesis | up to 4 weeks
  protein synthesis is evaluated in muscle biopsy tissue

SECONDARY OUTCOMES:
body composition is evaluated using DEXA | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University